CLINICAL TRIAL: NCT00005081
Title: Phase II Trial of BCNU Plus O6-Benzylguanine in the Treatment of Patients With Recurrent or Progressive Cerebral Anaplastic Gliomas
Brief Title: Carmustine Plus O6-benzylguanine in Treating Patients With Recurrent or Progressive Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0059; DUMC-0059-00-1; DUMC-T98-0059; NCI-T98-0059; CDR0000067688
Record Dates: First submitted 2000-04-06; First posted 2004-05-03 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Glioma; Gliosarcoma | interventions — O(6)-benzylguanine; Carmustine

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: carmustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining carmustine and O6-benzylguanine in treating patients who have recurrent or progressive glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the activity of carmustine and O6-benzylguanine in patients with recurrent or progressive glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma resistant to nitrosourea. II. Determine the toxic effects of this regimen in these patients.

OUTLINE: Patients receive O6-benzylguanine IV over 1 hour, followed 1 hour later by carmustine IV over 1 hour on day 1. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 18-32 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or progressive glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma Resistant to nitrosourea (defined as progressive or recurrent disease within 8 weeks of receiving nitrosourea) Measurable residual disease by MRI or CT scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin greater than 10 g/dL Hepatic: Bilirubin normal SGOT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL BUN no greater than 25 mg/dL Pulmonary: DLCO greater than 80% predicted Other: Not pregnant or nursing Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy At least 6 weeks since prior nitrosourea, procarbazine, or mitomycin and recovered No prior nitrosourea greater than 1,200 mg/m2 Endocrine therapy: Concurrent stable dose corticosteroids allowed if on for at least two weeks prior to study Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States